CLINICAL TRIAL: NCT00002807
Title: A Phase III Randomized Trial Comparing TAH BSO Versus TAH BSO Plus Adjuvant Pelvic Irradiation in Intermediate Risk Carcinoma of the Endometrium
Brief Title: Radiation or Observation Only in Endometrial Cancer Who Have Undergone Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN5; CAN-NCIC-EN5 (Other: PDQ); NCI-V96-0945 (Other Grant/Funding Number: NCI); CDR0000064915 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Endometrial Cancer
Keywords: stage I endometrial carcinoma; stage II endometrial carcinoma; endometrial adenocarcinoma; endometrial adenosquamous cell carcinoma; endometrial papillary carcinoma; endometrial clear cell carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Observation (No Intervention)
- Radiation (Experimental): Post-operative pelvic radiation therapy (45 Gy in 25 fractions over 5 weeks)
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — 45 Gy in 25 fractions over 5 weeks
  Arms: Radiation

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage cancer cells. It is not yet known whether radiation therapy is more effective than observation only after sugery in treating endometrial cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared to observation only in treating patients with stage I or stage II endometrial cancer who have undergone hysterectomy and oophorectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival in patients with intermediate-risk endometrial cancer treated with pelvic radiotherapy vs observation after laparoscopically-assisted vaginal hysterectomy or total abdominal hysterectomy and bilateral salpingo-oophorectomy.
* Compare the time to locoregional recurrence (i.e., in the vaginal mucosa or elsewhere in the central pelvic area or lateral pelvic walls) in patients treated with these regimens.
* Compare the duration of ultimate pelvic control and event-free survival in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare sexual health issues in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center, tumor grade (1 vs 2 vs 3), surgical staging (yes vs no), and sexual health assessment (yes vs no).

Patients undergo laparoscopic-assisted vaginal hysterectomy or total abdominal hysterectomy and bilateral salpingo-oophorectomy. After surgery, patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo observation alone.
* Arm II: Beginning within 12 weeks (preferably within 6-8 weeks) after surgery, patients undergo radiotherapy 5 days a week for 5 weeks in the absence of disease progression or unacceptable toxicity. Protocol-defined brachytherapy is allowed.

Quality of life is assessed at baseline; at 16-18 weeks after surgery (arm I) or 5 and 9 weeks after initiating radiotherapy (arm II); and then at 6, 12, 18, 24, 36, 48, and 60 months.

Patients are followed every 3 months for 2 years, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma or adenosquamous cell carcinoma of the endometrium

  * Intermediate-risk of recurrence after laparoscopically-assisted vaginal hysterectomy (with or without laparoscopic staging) or total abdominal hysterectomy and bilateral salpingo-oophorectomy
  * Postoperative pathologic stage IA/IB (grade 3), stage IC (grade 1-3), or stage IIA (all grades)
* Patients with more than 50% myometrial invasion (grade 1 or 2) or less than 50% myometrial invasion (grade 3) but with positive peritoneal cytology also eligible

  * Patients whose sole criterion for increased risk is positive peritoneal cytology are not eligible
* No pathologically involved lymph nodes if staging procedure performed
* Stage I papillary serous or clear cell endometrial cancer allowed

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0-3

Life expectancy:

* At least 3 years

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Not specified

Renal:

* Creatinine less than 2 times upper limit of normal
* No serious renal disease that would preclude radiotherapy

Cardiovascular:

* No serious cardiovascular disease that would preclude radiotherapy

Other:

* No history of inflammatory bowel disease such as ulcerative colitis
* No other malignancy within past 5 years except curatively treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, colon cancer, or thyroid cancer
* No psychiatric or addictive disorder that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No prior anticancer hormonal therapy
* No concurrent progestogens

Radiotherapy:

* No prior pelvic irradiation
* No prior or other concurrent vaginal intracavitary radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No prior anticancer therapy
* No other concurrent anticancer therapy

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 1996-07-04 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2009-12-21 (Actual)

PRIMARY OUTCOMES:
Survival (combined with the ASTEC trial) | 2009

SECONDARY OUTCOMES:
Progression-free survival | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Himu R. Lukka, MD, Study Chair — Margaret and Charles Juravinski Cancer Centre; Timothy J. Whelan, MD, Study Chair — Margaret and Charles Juravinski Cancer Centre
Locations (25):
- St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota, United States
- Royal Women's Hospital, Carlton, Victoria, Australia
- Canada (23):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Fraser Valley Cancer Centre at British Columbia Cancer Agency, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre at Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario, Kingston, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Humber River Regional Hospital - Weston, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] ASTEC/EN.5 Study Group; Blake P, Swart AM, Orton J, Kitchener H, Whelan T, Lukka H, Eisenhauer E, Bacon M, Tu D, Parmar MK, Amos C, Murray C, Qian W. Adjuvant external beam radiotherapy in the treatment of endometrial cancer (MRC ASTEC and NCIC CTG EN.5 randomised trials): pooled trial results, systematic review, and meta-analysis. Lancet. 2009 Jan 10;373(9658):137-46. doi: 10.1016/S0140-6736(08)61767-5. Epub 2008 Dec 16. PMID 19070891